CLINICAL TRIAL: NCT07044557
Title: MeDex: No Perioperative Dexamethasone in Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Akshitkumar MIstry, M.D., Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25.0244
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Perioperative treatment of newly diagnosed cancer patients with brain metastasis without dexamethasone. We will conduct a single-arm trial, assessing the safety and efficacy of brain metastasis resection without perioperative Dex. We will assess efficacy by noting presence of absence of lymphopenia. The participants will be followed until initiation of postoperative adjuvant cancer therapy for collection of primary and secondary endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Withholding perioperative dexamethasone (Experimental): The safety and feasibility of withholding perioperative dexamethasone (Dex) in newly diagnosed cancer patients undergoing resection of brain metastases (BMs). The primary question is not comparative efficacy, but rather whether it is safe to forgo Dex in this patient population.
  Interventions: Other: Withholding perioperative Dexamethasone

INTERVENTIONS:
Other: Withholding perioperative Dexamethasone — Patients will not receive perioperative Dex before, during, and up to 3 weeks after surgery.

SUMMARY:
Perioperative treatment of newly diagnosed cancer patients with brain metastasis without dexamethasone (Dex).

DETAILED DESCRIPTION:
This is a single-arm trial, assessing the safety and efficacy of brain metastasis resection without perioperative Dex in a maximum of 35 patients screened and enrolled in our emergency room and clinics. Investigators will assess efficacy by noting presence of absence of lymphopenia. The patients will be followed until initiation of postoperative adjuvant cancer therapy for collection of primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. New brain tumor(s) on imaging
2. Visceral mass(es) suspicious or confirmed for neoplasm

   a. Patients with lung mass suspicious for primary lung cancer and no prior diagnosis must undergo biopsy of the lung mass prior to resection of brain metastasis(es) to exclude histology (i.e., small cell lung carcinoma) that would not benefit from resection
3. No contraindications for craniotomy
4. Age ≥ 18 years
5. ECOG performance status ≤ 2 (i.e., ambulatory > 50% of waking hours)
6. Midline shift on MRI ≤ 10 mm
7. Craniotomy planned to resect >75% of the enhancing mass (surgeon's judgment)

Exclusion Criteria:

1. Presence of BMs not eligible for resection that are each > 2 cm in any one dimension
2. >4 BMs not eligible for resection that are each 2 cm in any one dimension
3. Treatment with laser interstitial thermal therapy (LITT)
4. High concern for primary CNS lymphoma
5. Diagnosis of small cell lung carcinoma
6. Any receipt of Dex
7. Steroid use in the past month
8. A condition that requires steroids
9. Stage 4 chronic kidney disease (GFR<30)
10. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dexamethasone Rescue Need | 4 weeks post operative (+-) 2 weeks
  Initiation of dexamethasone after enrollment up to 3 weeks after surgery.

SECONDARY OUTCOMES:
Immunosuppression Assessment | 4 weeks post operative (+-) 2 weeks
  Presence of absence of lymphopenia prior to adjuvant cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Akshitkumar Mistry, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States